CLINICAL TRIAL: NCT00658684
Title: An Open-Label, Multicenter, Long Term Study to Evaluate the Safety, Tolerability and Efficacy of Fesoterodine in Patients With Overactive Bladder.
Brief Title: Long Term Study To Evaluate the Safety, Tolerability and Efficacy of Fesoterodine for Overactive Bladder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0221006; A0221006
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fesoterodine fumarate (Experimental)
  Interventions: Drug: fesoterodine fumarate

INTERVENTIONS:
Drug: fesoterodine fumarate — 4 mg tablets OD for 4 weeks, then either 4 mg or 8 mg tablets OD for 48 weeks

SUMMARY:
To assess the long term safety, tolerability and efficacy of fesoterodine in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Adult OAB patients who present with OAB symptoms, including micturitions >= 8 per day and urinary urgency episodes >=1 per day.

Exclusion Criteria:

* Patient has known hypersensitivity to the active substance (fesoterodine fumarate) or to peanut or soya or any of the excipients.
* Patient has a known neurological disease influencing bladder function.
* Patient has a complication of lower urinary tract pathology potentially responsible for urgency or incontinence, clinically relevant bladder outlet obstruction or pelvic organ prolapse.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - Pfizer Investigational Site, Inegeku, Chibashi, Chiba
  - Pfizer Investigational Site, Akashi-shi, Hyōgo
  - Pfizer Investigational Site, Amagasaki-shi, Hyōgo
  - Pfizer Investigational Site, Chuou-ku, Koube-shi, Hyōgo
  - Pfizer Investigational Site, Kaibara-cho, Tanba-shi, Hyōgo
  - Pfizer Investigational Site, Nishinomiya-shi, Hyōgo
  - Pfizer Investigational Site, Kawasakishi, Kanagawa
  - Pfizer Investigational Site, Sagamihara-shi, Kanagawa
  - Pfizer Investigational Site, Nara, Nara
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Shibuya-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221006&StudyName=Long%20Term%20Study%20To%20Evaluate%20the%20Safety%2C%20Tolerability%20and%20Efficacy%20of%20Fesoterodine%20for%20Overactive%20Bladder.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 12 centers in Japan.
Pre-assignment Details: After screening, eligible subjects entered a run-in phase during which they completed a 3-day micturition diary for 3 consecutive days in 7 days prior to Baseline visit. At Baseline visit, the diary data and screening laboratory data were checked against the entry criteria to identify subjects eligible for study participation.
Groups:
- Total: All subjects
- 4 mg: Remained on a dose of fesoterodine 4 mg for the entire treatment period (subjects who remained on a dose of 4 mg)
- 4 mg > 8 mg > 4 mg: Increased to fesoterodine 8 mg at Week 4 and reduced to 4 mg at Week 8 (subjects whose dose was increased to 8 mg and then reduced to 4 mg)
- 4 mg > 8 mg: Increased to fesoterodine 8 mg at Week 4 and remained on a dose of 8 mg after Week 4 (subjects whose dose was increased to 8 mg and maintained)
Period: Overall Study
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Started | 152 | 99 | 25 | 28
Completed | 133 | 84 | 22 | 27
Not Completed | 19 | 15 | 3 | 1
Not completed — Adverse Event | 10 | 8 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg | Total
Number analyzed (Participants) | 99 | 25 | 28 | 152
Age Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.1) | 54.7 (10.5) | 57.0 (11.7) | 52.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 21 | 24 | 133
  Male | 11 | 4 | 4 | 19

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4, 8, 28 and 52
Description: The number of UUI episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean number of UUI episodes per 24 hours was calculated as the total number of UUI episodes for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: Of the efficacy analysis set, the subjects whose mean number of UUI episodes per 24 hours at baseline was greater than 0 were analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using last observation carried forward (LOCF) were analyzed. (n=number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 101 | 60 | 17 | 24
Number of episodes
  Baseline (n=101, 60, 17, 24) | 1.6 (1.48) | 1.4 (1.23) | 1.7 (1.24) | 2.1 (2.04)
  Week 4 (n=101, 60, 17, 24) | -0.86 (1.104) | -0.99 (1.117) | -0.73 (1.281) | -0.63 (0.918)
  Week 8 (n=100, 59, 17, 24) | -1.15 (1.293) | -1.16 (1.173) | -1.31 (1.450) | -1.00 (1.491)
  Week 28 (n=95, 56, 16, 23) | -1.28 (1.282) | -1.24 (1.185) | -1.25 (1.518) | -1.41 (1.385)
  Week 52 (n= 92, 54, 15, 23) | -1.34 (1.553) | -1.23 (1.228) | -1.18 (1.661) | -1.71 (2.097)
  Week 52 (LOCF) (n=101, 60, 17, 24) | -1.35 (1.521) | -1.19 (1.176) | -1.22 (1.568) | -1.82 (2.120)

2. Secondary Outcome: Change From Baseline in Mean Number of Micturitions at Week 4, 8, 28 and 52
Description: The number of micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean number of micturitions per 24 hours was calculated as the total number of micturitions for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: The efficacy analysis set (those who took at least one dose of study drug and contributed data to baseline and at least one valid post-baseline efficacy assessment) was analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using LOCF were also analyzed. (n=number of anlyzable subjects)
Measure: Mean (Standard Deviation); unit: Number of micturitions
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Number of micturitions
  Baseline (n=150, 97, 25, 28) | 11.3 (2.85) | 11.0 (2.69) | 11.2 (2.71) | 12.3 (3.31)
  Week 4 (n=150, 97, 25, 28) | -1.42 (1.855) | -1.73 (1.899) | -1.28 (1.403) | -0.45 (1.757)
  Week 8 (n=148, 95, 25, 28) | -2.11 (1.946) | -2.03 (1.897) | -1.81 (2.035) | -2.63 (2.005)
  Week 28 (n=137, 87, 23, 27) | -2.33 (2.338) | -2.18 (2.351) | -2.06 (2.260) | -3.02 (2.315)
  Week 52 (n=133, 84, 22, 27) | -2.63 (2.220) | -2.48 (2.02) | -2.21 (2.196) | -3.44 (2.683)
  Week 52 (LOCF) (n=150, 97, 25, 28) | -2.49 (2.172) | -2.35 (1.970) | -2.04 (2.135) | -3.36 (2.673)

3. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Week 4, 8, 28 and 52
Description: The number of urgency episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean number of urgency episodes per 24 hours was calculated as the total number of urgency episodes for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: The efficacy analysis set (those who took at least one dose of study drug and contributed data to baseline and at least one valid post-baseline efficacy assessment) was analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using LOCF were also analyzed. (n=number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Number of episodes
  Baseline (n=150, 97, 25, 28) | 4.5 (3.40) | 3.9 (3.31) | 6.2 (3.72) | 5.1 (2.87)
  Week 4 (n=150, 97, 25, 28) | -1.69 (2.009) | -1.77 (1.856) | -1.75 (2.572) | -1.37 (2.001)
  Week 8 (n=148, 95, 25, 28) | -2.44 (2.194) | -2.32 (1.881) | -2.59 (2.940) | -2.70 (2.463)
  Week 28 (n=137, 87, 23, 27) | -2.54 (2.597) | -2.41 (1.855) | -3.12 (3.304) | -2.46 (3.780)
  Week 52 (n=133, 84, 22, 27) | -2.76 (2.901) | -2.55 (2.579) | -2.80 (3.193) | -3.37 (3.565)
  Week 52 (LOCF) (n=150, 97, 25, 28) | -2.61 (2.885) | -2.30 (2.531) | -2.93 (3.319) | -3.40 (3.504)

4. Secondary Outcome: Change From Baseline in Mean Incontinence Episodes Per 24 Hours at Week 4, 8, 28 and 52
Description: The number of incontinence episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean number of incontinence episodes per 24 hours was calculated as the total number of incontinence episodes for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: Of the efficacy analysis set, the subjects whose mean number of incontinence episodes per 24 hours at baseline was greater than 0 were analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using LOCF were also analyzed. (n= number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 103 | 62 | 17 | 24
Number of episodes
  Baseilne (n=103, 62, 17,24) | 1.8 (1.74) | 1.6 (1.34) | 1.8 (1.33) | 2.5 (2.63)
  Week 4 (n=103, 62, 17,24) | -0.84 (1.140) | -0.99 (1.166) | -0.80 (1.225) | -0.49 (0.963)
  Week 8 (n=102, 61, 17, 24) | -1.23 (1.354) | -1.16 (1.272) | -1.43 (1.504) | -1.28 (1.486)
  Week 28 (n= 97, 58, 16, 23) | -1.39 (1.476) | -1.26 (1.322) | -1.31 (1.542) | -1.77 (1.779)
  Week 52 (n=94, 56, 15, 23) | -1.37 (1.589) | -1.26 (1.331) | -1.16 (1.847) | -1.75 (1.962)
  Week 52 (LOCF) (n=103, 62, 17,24) | -1.38 (1.557) | -1.24 (1.282) | -1.20 (1.740) | -1.86 (1.990)

5. Secondary Outcome: Change From Baseline in Number of Nighttime Micturitions Per 24 Hours at Week 4, 8, 28 and 52
Description: The number of nighttime micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean number of nighttime micturitions per 24 hours was calculated as the total number of nighttime micturitions for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: Of the efficacy analysis set, the subjects whose mean number of nighttime micturitions per 24 hours at baseline was greater than 0 were analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using LOCF were also analyzed. (n=number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: Number of micturitions
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 116 | 69 | 23 | 24
Number of micturitions
  Baseline (n=116, 69, 23, 24) | 1.4 (1.04) | 1.2 (1.04) | 1.6 (0.93) | 1.6 (1.05)
  Week 4 (n=116, 69, 23, 24) | -0.31 (0.727) | -0.34 (0.752) | -0.45 (0.556) | -0.08 (0.776)
  Week 8 (n=115, 68, 23, 24) | -0.43 (0.797) | -0.33 (0.812) | -0.55 (0.845) | -0.60 (0.688)
  Week 28 (n=106, 62, 21, 23) | -0.47 (0.752) | -0.36 (0.788) | -0.56 (0.694) | -0.71 (0.661)
  Week 52 (n=103, 60, 20, 23) | -0.57 (0.807) | -0.46 (0.904) | -0.68 (0.546) | -0.75 (0.698)
  Week 52 (LOCF) (n=116, 69, 23, 24) | -0.50 (0.826) | -0.38 (0.908) | -0.62 (0.614) | -0.71 (0.718)

6. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Week 4, 8, 28 and 52
Description: Voided volume per micturition was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  The mean voided volume per micturitions was calculated as the total voided volume for valid diary days divided by the total number of valid diary days collected at that visit.
  Change: mean at Week 4, 8, 28 and 52 minus mean at Baseline
Time Frame: Week 4, 8, 28 and 52
Population: The efficacy analysis set (those who took at least one dose of study drug and contributed data to baseline and at least one valid post-baseline efficacy assessment) was analyzed. Observed values were used for the analyses. Only at Week 52, the imputed data for missing values by using LOCF were analyzed. (n=number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
mL
  Baseline (n=150, 97, 25, 28) | 158.1 (48.09) | 162.8 (48.78) | 156.1 (42.75) | 143.6 (48.73)
  Week 4 (n=150, 97, 25, 28) | 16.67 (41.908) | 20.58 (44.357) | 12.18 (43.399) | 7.16 (29.231)
  Week 8 (n=148, 95, 25, 28) | 22.34 (51.339) | 21.86 (58.194) | 23.00 (35.061) | 23.37 (38.273)
  Week 28 (n=137, 87, 23, 27) | 32.59 (46.389) | 31.98 (50.365) | 40.20 (41.613) | 28.10 (36.431)
  Week 52 (n=133, 84, 22, 27) | 35.92 (44.007) | 40.21 (47.646) | 33.02 (40.772) | 24.95 (32.414)
  Week 52 (LOCF) (n=150, 97, 25, 28) | 33.42 (45.175) | 37.08 (49.276) | 28.22 (40.693) | 25.38 (31.890)

7. Secondary Outcome: Change From Baseline in Score of King's Health Questionnaire (KHQ) at Week 28 and 52
Description: KHQ was used to assess the impact of bladder problems on quality of life. The scores ranged from 0 to 100, where 0=best outcome/response and 100=worst outcome/response. A negative change indicates improvement.
  KHQ consists of the following domains:
  * General health perceptions (GHP)
  * Impact on life
  * Role limitations
  * Physical limitations
  * Social limitations
  * Personal relationships (PR)
  * Emotions
  * Sleep/energy
  * Incontinence severity measures (ISM)
  Change: mean at Week 28 and 52 minus mean at Baseline
Time Frame: Week 28 and 52
Population: The efficacy analysis set (those who took at least one dose of study drug and contributed data to baseline and at least one valid post-baseline efficacy assessment) was analyzed. Observed values were used for the analyses. (n=number of analyzable subjects)
Measure: Mean (Standard Deviation); unit: Scores on a ascle
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Scores on a ascle
  GHP: Baseline (n=150, 97, 25, 28) | 37.5 (21.63) | 37.1 (21.38) | 37.0 (24.07) | 39.3 (20.89)
  GHP: Week 28 (n=137, 87, 23, 27) | -2.19 (24.903) | -0.57 (26.131) | 0.00 (22.613) | -9.26 (22.088)
  GHP: Week 52 (n=134, 85, 22, 27) | -5.22 (22.751) | -5.88 (23.981) | -5.68 (21.729) | -2.78 (20.016)
  Impact on life: Baseline (n=150, 97, 25, 28) | 64.0 (23.97) | 61.2 (21.88) | 68.0 (31.15) | 70.2 (22.84)
  Impact on life: Week 28 (n=137, 87, 23, 27) | -32.85 (27.112) | -32.18 (24.084) | -37.68 (33.791) | -30.86 (30.559)
  Impact on life: Week 52 (n=134, 85, 22, 27) | -33.08 (29.333) | -32.94 (26.970) | -31.82 (33.297) | -34.57 (33.945)
  Role limitations: Baseline (n=150, 97, 25, 28) | 47.9 (24.75) | 46.0 (23.05) | 52.0 (30.55) | 50.6 (25.04)
  Role limitations: Week 28 (n=137, 87, 23, 27) | -28.10 (24.733) | -28.16 (22.777) | -33.33 (28.427) | -23.46 (27.448)
  Role limitations: Week 52 (n=134, 85, 22, 27) | -29.85 (26.732) | -30.98 (26.371) | -31.06 (28.310) | -25.31 (27.100)
  Physical limitations: Baseline (n=150, 97, 25, 28 | 51.9 (26.93) | 49.8 (26.73) | 54.0 (29.38) | 57.1 (25.43)
  Physical limitations: Week 28 (n=137, 87, 23, 27) | -27.25 (26.031) | -26.63 (25.727) | -31.16 (29.432) | -25.93 (24.605)
  Physical limitations: Week 52 (n=134, 85, 22, 27) | -30.10 (25.071) | -32.16 (24.504) | -28.03 (25.915) | -25.31 (26.300)
  Social limitations: Baseline (n=150, 97, 25, 28) | 30.3 (24.36) | 27.5 (23.38) | 31.1 (25.86) | 39.3 (25.03)
  Social limitations: Week 28 (n=137, 87, 23, 27) | -19.63 (19.410) | -17.37 (19.241) | -22.71 (19.955) | -24.28 (19.006)
  Social limitations: Week 52 (n=134, 85, 22, 27) | -22.35 (22.661) | -20.72 (22.245) | -24.75 (21.668) | -25.51 (25.000)
  PR: Baseline (n=124, 82, 18, 24) | 19.5 (22.46) | 17.3 (20.86) | 16.7 (22.87) | 29.2 (25.66)
  PR: Week 28 (n=110, 71, 16, 23) | -13.18 (18.354) | -11.74 (18.558) | -10.42 (17.078) | -19.57 (17.875)
  PR: Week 52 (n=109, 70, 16, 23) | -14.68 (19.342) | -13.57 (19.514) | -12.50 (17.743) | -19.57 (19.881)
  Emotions: Baseline (n=150, 97, 25, 28) | 51.2 (28.38) | 49.1 (27.49) | 52.0 (32.19) | 57.5 (27.89)
  Emotions: Week 28 (n=137, 87, 23, 27) | -27.49 (24.219) | -27.84 (23.163) | -27.54 (26.137) | -26.34 (26.714)
  Emotions: Week 52 (n=134, 85, 22, 27) | -30.27 (26.434) | -32.42 (24.799) | -26.26 (28.595) | -26.75 (29.760)
  Sleep/energy: Baseline (n=150, 97, 25, 28) | 37.0 (27.44) | 33.2 (24.00) | 37.3 (29.77) | 50.0 (33.02)
  Sleep/energy: Week 28 (n=137, 87, 23, 27) | -18.61 (21.586) | -17.43 (19.998) | -18.12 (26.070) | -22.84 (22.715)
  Sleep/energy: Week 52 (n=134, 85, 22, 27) | -21.27 (23.338) | -20.59 (22.219) | -15.91 (22.700) | -27.78 (26.554)
  ISM: Baseline (n=150, 97, 25, 28) | 34.8 (20.39) | 32.6 (18.83) | 31.5 (18.51) | 45.7 (24.05)
  ISM: Week 28 (n=137, 87, 23, 27) | -16.25 (17.223) | -14.87 (16.541) | -16.81 (17.623) | -20.25 (18.990)
  ISM: Week 52 (n=134, 85, 22, 27) | -19.00 (19.199) | -18.43 (18.392) | -14.55 (19.370) | -24.44 (21.001)

8. Secondary Outcome: Change From Baseline in Score of Overactive Bladder Questionnaire (OAB-q) at Week 28 and 52
Description: OAB-q was used to assess the extent of subjects who had been botehred by selected bladder symptoms and to assess the effect on their health-related quality of life (HRQL). OAB-q consists of the symptom bother score(SBS), the HRQL total score and subscale scores (Coping, Concern, Sleep and Social). The SBS ranges from 0 to 100, where 0=minimal severity and 100=greatest severity (negative change indicates improvement). The HRQL scores range from 0 to 100, where 0=worst outcome and 100=best outcome (positive change indicates improvement).
  Change: mean at Week 28 and 52 minus mean at baseline
Time Frame: Week 28 and 52
Population: The efficacy analysis set (those who took at least one dose of study drug and contributed data to baseline and at least one valid post-baseline efficacy assessment) was analyzed. Observed values were used for the analyses. (n=analyzable subjects)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Scores on a scale
  SBS: Baseline (n=150, 97, 25, 28) | 42.7 (22.53) | 37.4 (19.74) | 45.2 (21.04) | 58.7 (25.55)
  SBS: Week 28 (n=137, 87, 23, 27) | -25.13 (19.835) | -22.30 (18.588) | -27.07 (16.231) | -32.59 (24.578)
  SBS: Week 52 (n=134, 85, 22, 27) | -25.24 (20.287) | -22.41 (17.616) | -21.25 (16.597) | -37.41 (26.206)
  HRQL-Total: Baseline (n=150, 97, 25, 28) | 70.7 (18.31) | 73.9 (16.66) | 72.2 (18.97) | 58.4 (18.64)
  HRQL-Total: Week 28 (n=137, 87, 23, 27) | 15.66 (14.711) | 14.26 (13.366) | 16.00 (14.787) | 19.88 (18.191)
  HRQL-Total: Week 52 (n=134, 85, 22, 27) | 16.92 (16.461) | 15.99 (14.717) | 13.35 (14.961) | 22.76 (21.365)
  HRQL-Coping: Baseline (n=150, 97, 25, 28) | 61.6 (26.07) | 65.6 (24.59) | 64.6 (26.49) | 45.1 (25.04)
  HRQL-Coping: Week 28 (n=137, 87, 23, 27) | 20.86 (20.008) | 19.66 (17.871) | 18.15 (18.605) | 27.04 (26.339)
  HRQL-Coping: Week 52 (n=134, 85, 22, 27) | 21.75 (23.773) | 20.91 (21.821) | 15.00 (18.127) | 29.91 (31.259)
  HRQL-Concern: Baseline (n=150, 97, 25, 28) | 71.0 (21.54) | 73.9 (19.70) | 72.5 (20.90) | 59.5 (24.98)
  HRQL-Concern: Week 28 (n=137, 87, 23, 27) | 18.48 (18.180) | 16.95 (17.142) | 21.24 (17.943) | 21.06 (21.515)
  HRQL-Concern: Week 52 (n=134, 85, 22, 27) | 19.77 (18.400) | 19.23 (16.946) | 16.49 (17.961) | 24.13 (22.669)
  HRQL-Sleep: Baseline (n=150, 97, 25, 28) | 66.5 (23.95) | 69.9 (22.30) | 65.8 (25.61) | 55.6 (25.45)
  HRQL-Sleep: Week 28 (n=137, 87, 23, 27) | 12.41 (21.808) | 11.13 (21.579) | 13.22 (19.313) | 15.85 (24.769)
  HRQL-Sleep: Week 52 (n=134, 85, 22, 27) | 14.90 (21.467) | 13.32 (19.629) | 13.09 (19.873) | 21.33 (27.197)
  HRQL-Social: Baseline (n=150, 97, 25, 28) | 89.2 (14.17) | 91.2 (12.31) | 90.6 (13.71) | 81.0 (17.81)
  HRQ- Social: Week 28 (n=137, 87, 23, 27) | 6.66 (11.461) | 5.01 (10.064) | 8.00 (13.156) | 10.81 (13.304)
  HRQL-Social: Week 52 (n=134, 85, 22, 27) | 7.22 (12.277) | 6.26 (10.537) | 6.55 (12.802) | 10.81 (16.222)

9. Secondary Outcome: The Number of Subjects Shifted in Patient Perception of Bladder Condition (PPBC) Responses From Baseilne to Week 28 and 52 Assessment and Its Percentage
Description: The number of subjects whose perception of bladder condition improved at least by one grade on PPBC from baseline at Week 28 and 52. The PPBC was rated on a 6-point scale as follows:
  1. no problems at all
  2. some very minor problems
  3. some minor problems
  4. some moderate problems
  5. severe problems
  6. many severe problems
Time Frame: Week 28 and 52
Population: as for outcome 7
Measure: Number; unit: Number of subjects
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Number of subjects
  Week 28 (n=137, 87, 23, 27) | 115 | 75 | 21 | 19
  Week 52 (n=134, 85, 22, 27) | 116 | 75 | 18 | 23

10. Secondary Outcome: Change From Baseline in Grade of PPBC at Week 28 and 52
Description: The PPBC assessment was rated on a 6-point scale as follows:
  1. no problems at all
  2. some very minor problems
  3. some minor problems
  4. some moderate problems
  5. severe problems
  6. many severe problems
  Change: mean at Week 28 and 52 minus mean at baseline A negative change indicates improvement.
Time Frame: Week 28 and 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 150 | 97 | 25 | 28
Scores on a scale
  Baseline (n=150, 97, 25, 28) | 4.3 (0.51) | 4.2 (0.43) | 4.5 (0.65) | 4.4 (0.56)
  Week 28 (n=137, 87, 23, 27) | -1.66 (1.166) | -1.74 (1.094) | -1.83 (0.937) | -1.26 (1.483)
  Week 52 (n=134, 85, 22, 27) | -1.78 (1.141) | -1.85 (1.139) | -1.59 (1.054) | -1.70 (1.235)

11. Primary Outcome: Safety Measurement Based on Adverse Events (AEs), Vital Signs, Clinical Laboratory Test, 12-lead ECG and Residual Urine Volume
Description: The number of subjects who experienced AEs (all causality and treatment-related ) based on safety assessment during the study were summarized. The severity and seriousness of treatment-emergent AEs as well as discontinuations, dose reductions and temporary discontinuations (DR/TD) due to treatment-emergent AEs were also summarized.
Time Frame: 52 Weeks
Population: The safety analysis set (all subjects who took at least one dose of study drug) was analyzed.
Measure: Number; unit: Number of subjects
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Number analyzed (Participants) | 152 | 99 | 25 | 28
Number of subjects
  All-causality AEs | 138 | 91 | 25 | 22
  Treatment-related AEs | 102 | 61 | 25 | 16
  Serious AEs | 1 | 1 | 0 | 0
  Severe AEs | 0 | 0 | 0 | 0
  Discontinuations due to all-causlity AEs | 10 | 8 | 2 | 0
  Discontinuations due to treatment-related AEs | 7 | 6 | 1 | 0
  DR/TD due to all-causality AEs | 30 | 6 | 23 | 1
  DR/TD due to treatment-related AEs | 23 | 0 | 23 | 0

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Total | 4 mg | 4 mg > 8 mg > 4 mg | 4 mg > 8 mg
Serious Adverse Events (participants affected / at risk) | 1/152 | 1/99 | 0/25 | 0/28
Other Adverse Events (participants affected / at risk) | 138/152 | 91/99 | 25/25 | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=152) | 4 mg (N=99) | 4 mg > 8 mg > 4 mg (N=25) | 4 mg > 8 mg (N=28)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=152) | 4 mg (N=99) | 4 mg > 8 mg > 4 mg (N=25) | 4 mg > 8 mg (N=28)
Vertigo (Ear and labyrinth disorders) | 3 | 2 | 0 | 1
Vision blurred (Eye disorders) | 3 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 1 | 1
Constipation (Gastrointestinal disorders) | 20 | 11 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 5 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 77 | 43 | 21 | 13
Gastritis (Gastrointestinal disorders) | 9 | 8 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 2 | 1
Periodontitis (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 3 | 0 | 1
Cystitis (Infections and infestations) | 12 | 8 | 1 | 3
Gastroenteritis (Infections and infestations) | 3 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 50 | 35 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12 | 1 | 3
Dizziness (Nervous system disorders) | 6 | 3 | 2 | 1
Headache (Nervous system disorders) | 5 | 5 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 6 | 2 | 3 | 1
Residual urine (Renal and urinary disorders) | 3 | 1 | 2 | 0
Urine flow decreased (Renal and urinary disorders) | 4 | 1 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.